CLINICAL TRIAL: NCT04611893
Title: Monitoring of NOAC Therapy: Standardizing Reference Intervals
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Specialist Resident, Chinese University of Hong Kong
Other Study IDs: Crec 2020.376
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; Stroke, Acute; Stroke Syndrome; Ischemic
Keywords: stroke; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests for haemoglobin level, platelet count, activated partial thromboplastin time (aPTT), prothrombin time (PT), international normalized ratio (INR), creatinine clearance (by Cockcroft-Gault formula), alanine aminotransferase, alkaline phosphatase, bilirubin, modified thrombin time (dabigatran users), factor-Xa assay (for apixaban, rivaroxaban users) will be performed at the same time as blood taking for NOAC levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic stroke patient: Ischemic stroke patients who are on dabigatran, apixaban and rivaroxaban based on the above inclusion and exclusion criteria will be recruited from the Prince of Wales Hospital, either in-patient or out-patient clinic

SUMMARY:
This study is aimed to establish reference intervals of NOAC (dabigatran, apixaban and rivaroxaban) in ethnic Chinese patients.

DETAILED DESCRIPTION:
360 patients who are on dabigatran, apixaban and rivaroxaban based on the above inclusion and exclusion criteria will be recruited. After the informed consent, the patient will be needed for blood taking before and 2 hours after the medication (NOAC). The patient's demographic data and medical history will also be retreived from Central Medical Syetem too.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Chinese ONLY
2. 18 years old or above
3. Non-valvular atrial fibrillation
4. Duration of NOAC use at least 3 months
5. No changes in NOAC dosage or type within 3 months
6. Creatinine Clearance (by Cockcroft-Gault formula) >/=30mL/min

Exclusion Criteria:

1. Valvular atrial fibrillation or no atrial fibrillation
2. Recent haemorrhage or ischemia within 1 year
3. Active liver disease
4. Abnormal baseline clotting profile
5. Abnormal baseline thrombocytopenia or thrombocytosis
6. Thromboembolic tendency other than atrial fibrillation (e.g. antiphospholipid syndrome, protein C, S, anti-thrombin III deficiency)
7. Non-compliant patients, defined as missing any doses of NOAC in recent 1 month
8. Anticoagulation for disorders other than AF
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are on dabigatran, apixaban and rivaroxaban based on the above inclusion and exclusion criteria will be recruited from the Prince of Wales Hospital, either in-patient or out-patient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
NOAC level in blood | One week after the recruitment
  The NOAC level in blood before and after the medication

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Ming Bonaventure IP, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No